CLINICAL TRIAL: NCT03390881
Title: Assessment of the Validity of Breath Acetone Concentration as a Bio-marker of Instantaneous Energy Balance in Healthy Subjects
Brief Title: Use of Breath Acetone aa a Marker of Energy Balance
Acronym: ACEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Empa - Swiss Federal Laboratories for Materials Testing and Research, Zürich (Unknown)
Responsible Party: Principal Investigator, Luc Tappy, MD, MD, University of Lausanne
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-01740
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Fasting; Fed
Keywords: breath acetone; energy balance
MeSH Terms: conditions — Fasting; Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasting condition (Experimental): Effects of cumulated negative energy balance (fasting over 480 min) on breath acetone changes
  Interventions: Other: Fasting condition
- Sugar condition (Active Comparator): Effects of sugar consumption on breath acetone changes
  Interventions: Other: Sugar condition
- Fat condition (Active Comparator): Effects of fat consumption on breath acetone changes
  Interventions: Other: Fat condition

INTERVENTIONS:
Other: Fasting condition — Subjects will fast over the whole experimental period (480 min)
  Arms: Fasting condition
Other: Sugar condition — After a 2-h fasting state, subjects will ingest every hour a drink containing 70% carbohydrate, 15% fat and 15% protein and providing 1.5 X hourly resting energy requirement.
  Arms: Sugar condition
Other: Fat condition — After a 2-h fasting state, subjects will ingest every hour a drink containing 70% fat, 15% carbohydrate and 15% protein and providing 1.5 X hourly resting energy requirement.
  Arms: Fat condition

SUMMARY:
This study aims at assessing whether breath acetone concentration is a good bio-marker of instantaneous energy balance in healthy subjects.

DETAILED DESCRIPTION:
Each participant will be studied on three occasions, separated by 1-4 weeks. Each evaluation will consist in the same set of metabolic measurements, but will be performed fasting or during administration of a 70% fat or 70% carbohydrate liquid diet, according to a randomized order.

On each occasion, subjects will consume a standardized dinner the day before the experiment. They will remain fasted since 10 pm until the test day.

On the day of the experiments, one venous cannula will be inserted into a forearm vein for the collection of blood samples. An indirect calorimetry (measurement of respiratory gas exchanges using a ventilated canopy at rest, or a face mask during exercise) will be performed throughout the 6-hour test to measure energy expenditure and net substrate oxidation rate. Blood samples will be obtained every 60 min for the measurement of plasma glucose, insulin, free fatty acids, and beta-hydroxybutyrate concentrations. Breath samples will be also collected every 60 min (in 500 ml sampling bag) for the measurement of breath acetone concentration using a novel gas analyzer based on infrared laser spectroscopy.

Measurements will be done during 3 consecutive periods:

* 0-120 min: Fast + Rest: subjects will remain lying in bed in fasting conditions (negative energy balance).
* 120-360 min: Fed + Rest: subjects will remain in bed in a fasting state (C) or will receive every hour a liquid meal containing either 70% fat, 15% carbohydrate and 15% protein (Fat), or 70% carbohydrate, 15% fat and 15% protein (Sugar), corresponding to 1.5 X hourly resting energy requirement (positive energy balance).
* 360-480 min: Fed + Exercise: subjects will be transferred to an ergometric bicycle and will be asked to bike at a power output of 25 W [i.e. increasing total energy expenditure to ca. 2 time resting energy expenditure (negative energy balance)].

ELIGIBILITY:
Inclusion Criteria:

* BMI 19.5-29.9 kg/m2,
* Healthy

Exclusion Criteria:

* any known disease (with the exception of allergies);
* consumption of alcohol > 40 g/day;
* any current drug treatment (with the exception of contraceptive agents, antihistaminergic drugs for allergies, or multivitamin supplementations),
* history of lactose intolerance,
* history of exercise intolerance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Breath acetone | Every 60 min from 0 to 420 min
  Changes in breath acetone concentrations in conditions of positive vs. negative energy balance.

SECONDARY OUTCOMES:
Plasma parameters | Every 60 min from 0 to 420 min
  Relationship between breath acetone and plasma beta-hydroxybutyrate, glucose, free fatty acids and insulin concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — Department of Physiology, University of Lausanne, Switzerland
Locations (1):
- University of Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No